CLINICAL TRIAL: NCT00128596
Title: A Phase II Study of Trisenox (Arsenic Trioxide) in the Treatment of Unresectable Liver Cancer
Brief Title: Arsenic Trioxide in Treating Patients With Metastatic Liver Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: PCI-04-06060; CDR0000438662 (Registry Identifier: PDQ (Physician Data Query)); CTI-PCI-04-06060
Record Dates: First submitted 2005-08-08; First posted 2005-08-10 (Estimated); Last update posted 2017-04-27 (Actual); Status verified 2006-01

CONDITIONS: Liver Cancer
Keywords: adult primary hepatocellular carcinoma; advanced adult primary liver cancer; recurrent adult primary liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Arsenic Trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as arsenic trioxide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well arsenic trioxide works in treating patients with metastatic liver cancer that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of arsenic trioxide in patients with unresectable metastatic hepatocellular carcinoma.
* Determine the safety and tolerability of this drug in these patients.

OUTLINE: Patients receive a loading dose of arsenic trioxide IV over 1-2 hours once daily on days 1-5* in week 1 and then twice weekly in weeks 2-8. Courses repeat every 8 weeks in the absence of disease progression or unacceptable toxicity.

NOTE: *The 5-day loading dose is only administered during course 1.

After completion of study treatment, patients are followed at 30 days and then periodically for up to 2 years.

PROJECTED ACCRUAL: A total of 15-25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed hepatocellular carcinoma

  * Unresectable metastatic disease
* Ascites allowed provided it is minimal

PATIENT CHARACTERISTICS:

Age

* Over 18

Performance status

* 0-2

Life expectancy

* Not specified

Hematopoietic

* WBC > 2,500/mm^3
* Absolute neutrophil count > 1,500/mm^3
* Platelet count > 75,000/mm^3

Hepatic

* Bilirubin < 2.5 mg/dL
* AST < 2.5 times upper limit of normal

Renal

* Not specified

Cardiovascular

* QTc interval ≤ 460 msec AND potassium and magnesium normal

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile female patients must use effective double-method contraception for ≥ 4 weeks before, during, and for ≥ 4 weeks after completion of study treatment (during and for ≥ 4 weeks after completion of study treatment for male patients)
* No blood, ova, or sperm donation during study treatment
* Potassium > 4.0 mEq/dL
* Magnesium > 1.8 mg/dL

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent biologic therapy

Chemotherapy

* More than 4 weeks since prior and no other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 4 weeks since prior and no concurrent radiotherapy

Surgery

* Not specified

Other

* No other concurrent investigational agents

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2004-06; Primary Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Efficacy
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: T. Clark Gamblin, MD, Study Chair — UPMC Cancer Center at UPMC Presbyterian
Locations (1):
- UPMC Cancer Centers, Pittsburgh, Pennsylvania, United States